CLINICAL TRIAL: NCT04026997
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Dose Response of Oral CIN-102 in Adults With Idiopathic and Diabetic Gastroparesis
Brief Title: A Phase 2 Study of CIN-102 in Adults With Idiopathic and Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CinDome Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CIN-102-121
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): CIN-102 tablets by mouth twice daily for 14 days
  Interventions: Drug: CIN-102 Dose 1
- Cohort 1 - Placebo (Placebo Comparator): Placebo tablets by mouth twice daily for 14 days
  Interventions: Drug: Placebo
- Cohort 2 (Experimental): CIN-102 tablets by mouth twice daily for 14 days
  Interventions: Drug: CIN-102 Dose 2
- Cohort 2- Placebo (Placebo Comparator): Placebo tablets by mouth twice daily for 14 days
  Interventions: Drug: Placebo
- Cohort 3 (Experimental): CIN-102 tablets by mouth twice daily for 14 days
  Interventions: Drug: CIN-102 Dose 3
- Cohort 3- Placebo (Active Comparator): Placebo tablets by mouth twice daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-102 Dose 1 — CIN-102 Dose 1
  Arms: Cohort 1
Drug: CIN-102 Dose 2 — CIN-102 Dose 2
  Arms: Cohort 2
Drug: CIN-102 Dose 3 — CIN-102 Dose 3
  Arms: Cohort 3
Drug: Placebo — Placebo
  Arms: Cohort 1 - Placebo; Cohort 2- Placebo; Cohort 3- Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 2A study to evaluate safety, efficacy, PK, and dose response of oral CIN-102 in adults with idiopathic and diabetic gastroparesis. The study will assess three oral doses of CIN-102 versus placebo in three separate cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 70 years old.
* Current diagnosis of idiopathic or diabetic gastroparesis OR documented delayed gastric emptying.
* Presence of moderate to severe nausea.
* Body mass index (BMI) between 18 and 40 kg/m2, inclusive.
* Glycosylated hemoglobin level <11% at Screening.
* Willing to washout from ongoing treatment for gastroparesis.
* Able to understand and willing to comply with all study visits, procedures, restrictions, and provide written informed consent according to institutional and regulatory guidelines.

Exclusion Criteria:

* Other known disorder or treatment which could explain or contribute to symptoms of gastroparesis.
* Positive test for drugs of abuse at the screening or evaluation visits.
* Personal or family history of prolonged heart rate-corrected QT.
* History or evidence of clinically significant arrhythmia.
* History of gastrectomy, fundoplication, vagotomy, pyloroplasty, or bariatric surgery.
* Females who are pregnant, nursing, or planning on becoming pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in gastric emptying | Baseline (gathered on Days -10 to -3) to Day 14

SECONDARY OUTCOMES:
Change from baseline in gastric emptying terminal phase elimination half life | Baseline (gathered on Days -10 to -3) to Day 14
The change from baseline in ANMS GCSI-DD total scores | Day -14 to 14
The change from baseline in ANMS GCSI-DD subscale scores | Day -14 to 14

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Research Site 101, Chula Vista, California
  - Research Site 114, Jacksonville, Florida
  - Research Site 117, Miami, Florida
  - Research Site 118, Miami, Florida
  - Research Site 111, Atlanta, Georgia
  - Research Site 110, Kansas City, Kansas
  - Research Site 103, Louisville, Kentucky
  - Research Site 112, Marrero, Louisiana
  - Research Site 104, Monroe, Louisiana
  - Research Site 102, Boston, Massachusetts
  - Research Site 121, Omaha, Nebraska
  - Research Site 113, Las Vegas, Nevada
  - Research Site 109, Great Neck, New York
  - Research Site 120, Winston-Salem, North Carolina
  - Research Site 105, Tulsa, Oklahoma
  - Research Site 106, Philadelphia, Pennsylvania
  - Research Site 119, Summerville, South Carolina
  - Research Site 115, Rapid City, South Dakota
  - Research Site 107, Jackson, Tennessee